# Consent form for Participation in Research Study Entitled: "Alcohol Impaired Driving in the Natural Environment"

You are being invited to participate in a research study entitled "Alcohol Impaired Driving in the Natural Environment" sponsored by the University of Missouri and conducted under the direction of Dr. Denis M. McCarthy.

## **Purpose of the Study**

• This project is designed to examine the factors that influence the decision to drive after drinking alcohol or ride with a driver who has consumed alcohol. Approximately 40 people will participate in this study.

### Compensation

- For participating in this research study, you will be paid \$15 per hour for your session today (approximately 3 hours or \$45) and your closeout interview in two weeks (approximately 1 hour or \$15). You will also be paid \$30 per week for each of the two weeks you are in the study (\$60 for two weeks). You total compensation for the project will be about \$120, depending on the time it takes to complete your interview sessions.
- If you withdraw your participation once the study has begun, you will still receive payment commensurate with the time you spend here.
- Payment will be made in cash following completion of each session of the study.

## What Will Happen During the Study

- You will complete a number of questionnaire items pertaining to demographics, personality factors, substance use, attitudes towards drinking and driving, and other behaviors.
- You will complete several computer tasks designed to assess different components of cognitive functioning (e.g., working memory).
- You will complete a computerized gambles task requiring you to make choices between two hypothetical monetary outcomes.
- You will complete a computerized decision-making task requiring you to make hypothetical choices regarding transportation home after alcohol consumption.
- You will complete a detailed interview about alcohol use and alcohol-impaired driving.
- You will learn how to use the smartphone app and go over expectations of participation for the 2 weeks of assessment.
- Duration of participation in the first session of the study is approximately 3 hours.
- You will then complete 2 weeks of ambulatory assessment using a smartphone app that will assess attitudes and decision making regarding drinking and driving and other questions about drinking behavior.
- You will also be provided with a portable breathalyzer. You will be trained on how to use this device and will be
  asked to provide a breath sample to measure your alcohol consumption several times per day during the two
  weeks of the study.
- During this period, the smartphone will also collect information on your location and travel. This information will be combined with the other information you provide at the conclusion of the study.
- You will return to the lab for a second session lasting approximately 1 hour to complete an abridged interview about alcohol use and alcohol-impaired driving over the 2 week period and be debriefed.
- Total duration of participation in the study is 2 weeks.

#### **Potential Risks**

- Some of the questionnaire items related to substance abuse and risky behaviors may be sensitive in that they concern various personal problems that you might have experienced. Some items refer to illegal behaviors (e.g., drug use, arrests).
- All data that is collected in this project will be confidential. Only code numbers are used to identify records, and your name is not linked to this code number. Please do not put identifying information (name, social security

number, etc.) on study questionnaires. If any records are copied and collected by reviewers, these records can be reviewed without revealing identifying information about you.

- This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents or biosamples that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents or biosamples protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.
- The Certificate cannot be used to refuse a request for information that is needed for auditing or program evaluation by NIH, which is funding this project. You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

#### **Benefits**

• There are no benefits to you from participating in this study. The investigators may learn more about decision making strategies in substance use-related situations and how different participant characteristics are related to decision making as well as the potential use of mobile technology as an intervention method.

## **Voluntary Participation**

• Participation in this research is entirely voluntary. You may refuse to participate or withdraw at any time. You also have the right to refuse to answer any study question.

#### **Ouestions or Concerns**

If you have questions or problems related to this study, you may reach Dr. McCarthy at (573) 882-0426. You may contact the Campus Institutional Review Board at (573) 882-9585 or umcresearchirb@missouri.edu to ask about your rights or to report research-related problems.

## Consent

By signing below, you indicate that you have read the information in this consent form, and agree to be in the study. You also indicate that you have had the chance to ask questions about this study and that they have been answered by Dr. McCarthy or an associate. You understand that you may ask questions at any time during or following the study.

| are two copies of this form. You will keep one copy and return the other to the invest | |
|---|---|
| Participant Signature | Date |
| Witness Signature | Date |